CLINICAL TRIAL: NCT00811304
Title: Real-time Ultrasound Guided Labor Epidural Placement
Status: Withdrawn | Type: Observational
Why Stopped: We are unable to find a clip used to stabilize the epidural needle on the ultrasound probe to allow adequate epidural catheter placement.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Manuel C. Vallejo, MD / Associate Professor/University Faculty Member, Magee-Womens Hospital of UPMC
Other Study IDs: PRO08090016
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: Epidural Anesthesia
Keywords: ultrasound; labor epidural; failed epidural; outcome; Epidural insertion under realtime ultrasound guidance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- US group: All patients admitted to the labor and delivery suite who request an epidural for labor analgesia.

SUMMARY:
Specific Aim: The purpose of this study is to determine if labor epidural placement using real-time (concurrent) ultrasound guided placement is superior to the conventional "standard" epidural technique without the use of ultrasound at Magee-Womens Hospital.

Hypothesis: Ultrasound guided labor epidural placement in real-time will decrease the traditional epidural failure rate from 5% to 1%.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women of childbearing age (including children aged 14 years and above) who request epidural analgesia at Magee-Womens Hospital will be eligible to participate in the study.

Exclusion Criteria:

* Men will not be included.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All pregnant women in labor.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Failed epidural placement rate | From admission untill delivery

SECONDARY OUTCOMES:
The incidence of post dural puncture headache. | From insertion of epidural to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Manuel C Vallejo, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States